CLINICAL TRIAL: NCT00002222
Title: An Open Label Study of the Safety and Tolerability of Valganciclovir, an Oral Prodrug of Ganciclovir, for the Treatment of Cytomegalovirus Retinitis in Subjects With AIDS
Brief Title: A Study of Valganciclovir in the Treatment of Cytomegalovirus (CMV) Retinitis in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 268B
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-04

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Ganciclovir; Antiviral Agents; Drug Administration Schedule; Cytomegalovirus Retinitis; Prodrugs
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency | interventions — Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir

SUMMARY:
The purpose of this study is to see if valganciclovir is a safe treatment for CMV retinitis in patients who have been treated for this condition in the past. This study also examines the effectiveness of valganciclovir in preventing the recurrence of CMV retinitis.

DETAILED DESCRIPTION:
Patients receive valganciclovir twice a day for 21 days as induction therapy then daily as maintenance therapy. Patients are encouraged to remain on study for at least 3 months and will remain until common study closure.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed with caution:

* Acyclovir.
* Famciclovir.
* Valaciclovir.
* Imipenem-cilastatin.
* Myelosuppressive agents.

Patients must have:

* HIV infection with CMV retinitis.
* Minimum of 4 weeks prior treatment with ganciclovir, foscarnet, or cidofovir.
* Intraocular implant in either or both eyes, as long as CMV retinitis is active in one eye, upon approval by Roche.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms of conditions are excluded:

* Active extraocular CMV disease.
* Severe uncontrolled diarrhea or evidence of malabsorption.

Concurrent Medication:

Excluded:

* Foscarnet.
* Cidofovir.
* CMV hyperimmune globulin.
* Probenecid.

Patients with the following prior conditions are excluded:

* Ocular media opacities (corneal, aqueous, lens, or vitreous) preventing ophthalmologic retinal assessment.
* Simultaneous participation in another study (unless approved by Roche).

Required:

* A minimum of 4 weeks treatment with ganciclovir, foscarnet, or cidofovir.
* Approval required for prior use of investigational anti-CMV agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell AIDS Clinical Trials Unit, New York, New York, United States